CLINICAL TRIAL: NCT01177319
Title: Glutathione (GSH) In The Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Wellness Health & Pharmaceuticals, Inc. (Industry)
Responsible Party: Robert A. Hauser, MD, University of South Florida
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GSH
Record Dates: First submitted 2010-08-05; First posted 2010-08-09 (Estimated); Last update posted 2010-08-09 (Estimated); Status verified 2007-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Glutathione
MeSH Terms: conditions — Parkinson Disease | interventions — Glutathione

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Glutathione

SUMMARY:
This is an investigator initiated pilot study to examine the effects of GSH in PD. The goal of this study is to acquire some basic data regarding side effects and efficacy of this compound to determine if this is a possible treatment option that could be recommended to interested PD patients.

DETAILED DESCRIPTION:
Inclusion Criteria Idiopathic Parkinson's disease (2 of 3 of the cardinal symptoms, tremor, bradykinesia, rigidity) Mini Mental State Examination > 24 Anti-parkinsonian medications stable for one month Hoehn and Yahr II-IV

Exclusion Criteria Atypical parkinsonism History of seizure, drug addiction Use of typical neuroleptics Previous use of glutathione

Methods Study Design The study will be a parallel, double-blind, placebo controlled trial lasting one month with three glutathione injections per week. Glutathione will be supplied by Wellness Health and Pharmaceuticals in Birmingham, Alabama.

Drug Administration The drug or a placebo (1:1 ratio) will be administered intravenously at doses of 1400 mg on Monday, Wednesday and Friday of each week for a four-week period. The drug will be infused by an intravenous push over 10 minutes and will be diluted in 10cc of normal saline. Therefore, there will be twelve intravenous infusions of either GSH or placebo.

Randomization Randomization will be done by computerized techniques assigning either GSH or placebo for a four-week period.

Clinical Assessment Assessments will be done at baseline and at the end of one, two, three and four weeks during administration of drug and eight and twelve weeks after initiation of the trial. Patients will be asked to come to the clinic at approximately the same time of day for each infusion. The assessments will be done each Friday throughout the trial, once prior to the infusion of the glutathione/placebo and again one hour after the infusion. The following assessments will be done: Unified Parkinson's Disease Rating Scale, timed walking test, tapping test and clinical global assessment by both the physician and the patient. Patient diaries and the Parkinson's Disease Questionnaire, a quality of life measurement, will be done weekly. Patients will also be videotaped using a standard protocol. The treating physician will not be doing the assessments, all assessments will be done by a blinded investigator. Assessment forms can be found in the appendix.

Safety Assessments Vital signs - orthostatic, supine and standing blood pressure and pulse will be taken at baseline and again 10 minutes after the completion of each IV infusion.

ECG - an ECG will be done prior to the first infusion and approximately 10 minutes after the completion of each infusion.

Adverse Reactions Adverse events will be reported according to FDA regulations. Known side effects of intravenous GSH include difficulty administering the drug intravenously which can cause some discomfort or bruising at the site of needle entry, the formation of a small blood clot or swelling of the vein and surrounding tissues, bleeding from the puncture site and on rare occasions fainting or infection. Side effects of glutathione include fatigue and gastrointestinal disturbances. Adverse reactions will be assessed through an open patient inquiry at each visit. Patients will also be instructed to call the PI in the event of any adverse effects throughout the study.

Statistical Analysis The GSH and placebo groups will be compared on all measures using nonparametric statistics. Mann-Whitney U comparisons for independent samples will be used to detect differences between the two groups. Significance will be p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (2 of 3 of the cardinal symptoms:tremor, bradykinesia, rigidity)
* Mini Mental State Examination > 24
* Anti-parkinsonian medications stable for one month
* Hoehn and Yahr II-IV
* Age 18 and above

Exclusion Criteria:

* Atypical parkinsonism
* History of seizure, drug addiction
* Use of typical neuroleptics
* Previous use of glutathione

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Timed walking test
Tapping test

SECONDARY OUTCOMES:
CGI-clinical global assessment by both the physician and the patient
Patient diaries
Parkinson's Disease Questionnaire, a quality of life measurement

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Hauser, MD, MBA, Principal Investigator — University of South Florida
Locations (1):
- USF Parkinson's Disease and Movement Disorders Center, Tampa, Florida, United States